CLINICAL TRIAL: NCT03244319
Title: Explore the Efficacy and Safety of edoxabaN in Patients After Heart Valve Repair or Bioprosthetic vaLve Replacement (ENAVLE Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0506
Record Dates: First submitted 2017-08-06; First posted 2017-08-09 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-10

CONDITIONS: MV(Mitral Valve) Repair
MeSH Terms: interventions — edoxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edoxaban (Experimental)
  Interventions: Drug: Edoxaban
- Warfarin (Active Comparator)
  Interventions: Drug: Warfarin; Drug: parenteral anti-coagulant (UFH)

INTERVENTIONS:
Drug: Edoxaban — Patients who are randomly assigned to edoxaban group will be received 60mg qd or 30mg qd (creatinine clearance 30-49ml/min, body weight <60kg or concomitant use of certain P-glycoprotein inhibitors).
  Arms: Edoxaban
Drug: Warfarin — All patients who are assigned to VKA group, bridging with warfarin and UFH is mandatory until INR reach therapeutic target range (INR 2-3). Warfarin dose will be adjusted for maintain therapeutic range (INR 2-3) during follow up period.
  Arms: Warfarin
Drug: parenteral anti-coagulant (UFH) — parenteral anti-coagulant (UFH)
  Arms: Warfarin

SUMMARY:
1. objectives: The primary aim of ENAVLE is to explore the efficacy of edoxaban in patients with post mitral valve repair or bioprosthetic valve implantation
2. Primary / Secondary Endpoint

1) Efficacy Endpoint Evaluation: Occurrence of thromboembolic events and any thrombus at repaired ring or bioprosthetic valves detected by follow up echocardiography or 3D CT scan

2) Safety Endpoint Evaluation

* Dysfunction of treated valve caused by thrombosis on echocardiography or 3D CT scan
* Major or minor bleeding described in safety outcomes

DETAILED DESCRIPTION:
This study is an open labeled, parallel group, and randomization study. At 7 days after mitral valve repair, bioprosthetic MV or AV replacement surgery, warfarin or edoxaban will be started per oral route. All study patients started to receive bridging therapy with parenteral anti-coagulant (UFH) according to local practice before switching to warfarin or edoxaban. Among patients who take warfarin, international normalized ratio will be used to monitor the effectiveness of the anticoagulant warfarin as usual daily practice. All patients who are assigned to VKA group, bridging with warfarin and UFH is mandatory until INR reach therapeutic target range (INR 2-3). Warfarin dose will be adjusted for maintain therapeutic range (INR 2-3) during follow up period. Patients who are randomly assigned to edoxaban group will be received 60mg qd or 30mg qd ( creatinine clearance 30-49ml/min, body weight <60kg or concomitant use of certain P-glycoprotein inhibitors). Both drugs will be maintained for 3 months. During study period, all patients will be carefully monitored for thromboembolic events including valve dysfunction, and stroke or bleeding complication. At 3 months after surgery, 3 dimensional CT scan and echocardiography will be performed for detecting valvular dysfunction, any thrombus or bleeding in heart & lung.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-85 years with
* MV repair or Bioprosthetic MV or AV replacement
* Patients with written informed consent

Exclusion Criteria:

* Previous mechanical prosthetic heart valve replacement
* Patients who underwent TAVI
* Concomitant bioprosthetic valve replacement of mechanical tricuspid or pulmonary replacement at the time of the index valve replacement surgery
* Clinically relevant paravalvular leaks
* Previous history of endocarditis
* Complex congenital heart abnormality
* Acute coronary syndrome within one month
* Uncontrolled hypertension
* Previous history of hemorrhagic stroke
* At high risk for bleeding
* Active hepatitis or liver dysfunction (AST/ALT> 3times of upper normal limits)
* Creatinine clearance < 30ml/min
* Patients with a clear indication for long-term dual antiplatelet therapy
* Malignancy or radiation therapy within one month
* Treatment with selected drugs that my interact with edoxaban (specific P-gp inhibitors, ie. verapamil, quinidine; the short-term use of azithromycin, clarithromycin, erythromycin, oral itraconazole, oral ketoconazole)
* At of pregnancy or breastfeeding
* Known allergy to warfarin or edoxaban

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of thromboembolic event | 12 weeks
  Occurrence of thromboembolic events and any thrombus at repaired ring or bioprosthetic valves detected by follow up echocardiography or 3D CT scan

SECONDARY OUTCOMES:
Dysfunction of treated valve | 12 weeks
  Dysfunction of treated valve caused by thrombosis on echocardiography or 3D CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No